CLINICAL TRIAL: NCT04167423
Title: Thyroid Disease in Pregnancy and Its Impact on the Quality of Life
Brief Title: Mapping Health-related Quality of Life in Pregnant Women With Thyroid Disease.
Acronym: ThyPreQol2020
Status: Completed | Type: Observational
Sponsor: Value Outcomes Ltd. (Other)
Collaborators: Charles University, Czech Republic (Other); Institute of Health Information and Statistics of the Czech Republic (Other Government)
Responsible Party: Sponsor
Other Study IDs: ThyPreQol2020
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-04

CONDITIONS: Thyroid Diseases; Pregnancy Related; Quality of Life
Keywords: quality of life; EQ5D; ThyPRO-39; pregnancy; thyroid disease; thyrotropin; thyroxine; thyroid autoantibodies
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy: No thyroid disease in pregnancy defined as plasma TSH (thyrotropin), TPOAb (thyroperoxidase auto antibodies) or FT4 (free thyroxin) out of the ranges proposed by 2014 European Thyroid Association Guideline.
- hyperthyroidism: Thyroid disease in pregnancy defined as plasma TSH, or FT4 out of the ranges proposed by 2014 European Thyroid Association Guideline.
- hypothyroidism: Thyroid disease in pregnancy defined as plasma TSH, or FT4 out of the ranges proposed by 2014 European Thyroid Association Guideline.
- thyroid autoimmunity: Thyroid disease in pregnancy defined as plasma TPOAb out of the ranges proposed by 2014 European Thyroid Association Guideline.

SUMMARY:
Natural thyroid function changes during pregnancy. In up to tens of percent of pregnant women, these changes can lead to pathological fluctuations in hormone and antibody production. Although the effects on pregnancy and child development are well described, none has determined their influence on mother's emotional well-being and the quality of life.

At present, universal thyroid screening in pregnancy in the Czech Republic is not covered by health insurance. The aim of the project is to change this situation by providing quality of life estimate for the cost-effectiveness model.

This is a project of three specialized institutions aimed at mapping various aspects of the quality of life of pregnant women and describing the impact of thyroid disease on their lives. The project is a parallel study to a larger project Early screening for thyreopathy in pregnancy (CZ.03.2.63/0.0/0.0/15_039/0009643) supported by the European Fund Operational Programme Employment through the National screening centre. The data will be collected through online questionnaire from women enrolled in the Early screening for thyreopathy in pregnancy (CZ.03.2.63/0.0/0.0/15_039/0009643) who were screened for TSH, TPOAb and FT4.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* screened for laboratory signs of thyreopathy anytime during pregnancy
* willing/able to participate in online survey

Exclusion Criteria:

* women whose laboratory results were not available or inconclusive
* already participated in this survey by filling the online questionnaire
* not able to complete the entire questionnaire

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women who were screened for laboratory signs of thyreopathy during pregnancy.
  All screened women attending the study center will be proposed to participate.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Utility by five-dimensional five-level generic EuroQoL questionnaire (EQ5D 5L) | Immediately after the reception of laboratory results
  Health-related quality of life measured as EQ5D 5L questionnaire, score 1 is the best and -0,594 the worst

SECONDARY OUTCOMES:
Thyroid-Related Quality-of-Life Patient-Reported Outcome questionnaire short form (ThyPRO-39) | Immediately after the reception of laboratory results
  Health-related quality of life measured as ThyPRO-39 questionnaire, each domain scores between 0 and 100. The higher the score the worse the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tužil, MSc et Eng, Study Director — Value Outcomes Ltd. et First Medical Faculty at Charles University, Prague; Tomáš Doležal, MD et PhD, Study Chair — Value Outcomes Ltd.; Jana Bartáková, Ing et PhD, Study Chair — Value Outcomes Ltd. et First Medical Faculty at Charles University, Prague
Locations (7):
- Czechia (7):
  - MUDr. Milan Kučera. s.r.o., Kladno, Czech Republic
  - MUDr. Eva Novotná - FEMCARE s.r.o., Odolena Voda, Czech Republic
  - Mediva s.r.o., Prague, Czech Republic
  - MUDr.Tereza Šmrhová-Kovács, Tábor, Czech Republic
  - Nemocnice Havlíčkův Brod, Havlíčkův Brod
  - Všeobecná Fakultní Nemocnice, Prague
  - Oblastní nemocnice Příbram, a.s., Příbram

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tuzil J, Pilnackova BF, Watt T, Jiskra J, Koudelkova M, Novotna E, Tuzilova K, Dolezal T, Bartakova J. The Impact of Subclinical Hypothyroidism on the Quality of Life During Pregnancy: Mapping 5-Level Version of EQ-5D and ThyPRO-39. Value Health. 2023 Jul;26(7):1085-1097. doi: 10.1016/j.jval.2023.02.015. Epub 2023 Mar 5. PMID 36878311